CLINICAL TRIAL: NCT06877234
Title: An Exploratory Clinical Study on the Safety and Efficacy of the Ultrasonic Nerve Ablation System in the Treatment of Essential Hypertension
Brief Title: Safety and Efficacy of Modulated Ultrasound Renal Denervation for HTN（FIM）
Acronym: ModulationHTN1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Pulsecare Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MW-2301-T-01
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exploratory Clinical Study of the Ultrasound Nerve Ablation System (Experimental)
  Interventions: Procedure: Ultrasonic Nerve Ablation System

INTERVENTIONS:
Procedure: Ultrasonic Nerve Ablation System — Treatment of patients with essential hypertension using the ultrasonic nerve ablation system

SUMMARY:
This study is a prospective and exploratory clinical study, enrolling patients with essential hypertension. This study is planned to be conducted in 2 research institutions in China, and a total of 6 subjects are planned to be included. After the subjects sign the informed consent form (ICF) approved by the ethics committee, they will enter the screening procedure. Subjects who meet the inclusion criteria and do not meet any of the clinical exclusion criteria will be enrolled after undergoing renal artery CTA angiography.

All patients will undergo clinical evaluation and blood pressure measurement during the operation, at the time of discharge, and at 1 month, 2 months, 3 months, and 6 months after the operation.

It is recommended that the anti-hypertensive medications used before the operation should not be changed within 6 months after the operation for the cases. When the systolic blood pressure (SBP) is ≥ 180 mmHg or there are clinical symptoms caused by hypertension, the drug dosage should be increased as a priority, and then the anti-hypertensive medications should be adjusted. When the systolic blood pressure (SBP) is ≤ 120 mmHg or there are clinical symptoms caused by a decrease in blood pressure, the anti-hypertensive medications should be reduced.

ELIGIBILITY:
Inclusion Criteria:

Males or females aged 18 years old or above and 65 years old or below; Patients with essential hypertension; Patients who have been stably taking 2 or more antihypertensive drugs at conventional doses continuously for at least 4 weeks before enrollment, and whose blood pressure meets the following conditions: (1) The systolic blood pressure measured in the outpatient clinic is ≥150 mmHg and ≤180 mmHg, and the diastolic blood pressure measured in the outpatient clinic is ≥90 mmHg; (2) The systolic blood pressure measured by 24-hour ambulatory blood pressure monitoring (ABPM) is between 135 mmHg and 170 mmHg; The course of hypertension is more than 6 months; The diameter of the renal artery evaluated by renal artery CTA is ≥3 mm and the length is ≥20 mm; The patient or his/her legal representative signs a written informed consent form approved by the ethics committee before screening;

Exclusion Criteria:

Complicated with type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus (defined as plasma Hb1Ac ≥ 10.0%); Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m²; Previous implantation of an implantable cardioverter-defibrillator (ICD) or a pacemaker; History of myocardial infarction, syncope, intracerebral hemorrhage or cerebral infarction within 6 months before signing the informed consent form; Severe valvular heart stenosis; Any factors that may interfere with blood pressure measurement under any circumstances (for example, the patient has severe peripheral vascular disease, abdominal aortic aneurysm, hemorrhagic disorders such as thrombocytopenia, hemophilia, severe anemia); Patients with sleep apnea syndrome; Females who are pregnant or breastfeeding, or those who have a plan to conceive within the next year; Other serious organic diseases with an expected lifespan of less than 12 months; Participation in other clinical trials before screening and not yet completed;

Preoperative exclusion criteria based on CTA imaging:

a. Visual inspection shows that the diameter stenosis of the renal artery on either side > 50% or there is a renal artery aneurysm on either side; b. Previous history of renal artery interventional treatment; Other situations that the investigator deems unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The change in the average daytime systolic blood pressure two months after the operation | Two months after the operation
  That is, the difference between the average daytime (from 7:00 to 22:00) systolic blood pressure measured before the operation and the average daytime systolic blood pressure measured during the follow-up visit two months after the operation
Major adverse events within 30 days after the operation | Within 30 days after the operation
  Major adverse events include: all-cause mortality, renal complications, renal artery embolism events, complications of interventional treatment, hypertensive/hypotensive crises during hospitalization, and major cardiovascular and cerebrovascular complications.

SECONDARY OUTCOMES:
The changes in the average systolic blood pressure of ambulatory blood pressure during the daytime, at night and over 24 hours after the operation | 1 month, 3 months, 6 months after the operation
  Changes in the average systolic blood pressure of ambulatory blood pressure during the daytime, at night and over 24 hours after the operation (1 month, 3 months, 6 months) That is, the difference between the average systolic blood pressure of ambulatory blood pressure measured during the daytime (7:00-22:00), at night (22:00-7:00) and over 24 hours before the operation and the average systolic blood pressure of ambulatory blood pressure measured during the daytime, at night and over 24 hours during the postoperative follow-up.
Changes in the average diastolic blood pressure of ambulatory blood pressure during the daytime, at night and over 24 hours after the operation | 1 month, 2 months, 3 months, 6 months after the operation
  That is, the difference between the average diastolic blood pressure of ambulatory blood pressure measured during the daytime (7:00-22:00), at night (22:00-7:00) and over 24 hours before the operation, and the average diastolic blood pressure of ambulatory blood pressure measured during the daytime, at night and over 24 hours during the postoperative follow-up
The attainment rate of systolic blood pressure reaching the standard in the outpatient clinic after the operation | 1 month, 2 months, 3 months, 6 months after the operation
  That is, the proportion of subjects whose systolic blood pressure measured in the outpatient clinic during the postoperative follow-up is less than 140 mmHg.
The change in systolic blood pressure measured in the outpatient clinic after the operation | 1 month, 2 months, 3 months, 6 months after the operation
  That is, the difference between the systolic blood pressure measured in the outpatient clinic before the operation and the systolic blood pressure measured in the outpatient clinic during the postoperative follow-up
The average number of types of medications taken after the operation | 1 month, 2 months, 3 months, 6 months after the operation
  The change in the average number of types of medications taken during the postoperative follow-up period, compared with the antihypertensive medications taken before the operation.
The incidence rate of complications of interventional treatment | 1 month, 2 months, 3 months, 6 months after the operation
  It refers to the intraoperative or postoperative related complications that occur after the research device has completed the renal artery ultrasound ablation surgery, such as renal artery perforation, renal artery dissection, acute infection, etc
All-cause mortality rate | 1 month, 2 months, 3 months, 6 months after the operation
  Death caused by any reason as informed during the clinical follow-up
Cardiovascular and cerebrovascular complications | 1 month, 2 months, 3 months, 6 months after the operation
  It refers to myocardial infarction, any stroke event (including intracerebral hemorrhage and cerebral infarction), and any coronary revascularization
Renal complications | 1 month, 2 months, 3 months, 6 months after the operation
  Refers to eGFR <15 mL/min/1.73㎡, requirement for renal replacement therapy, or renal artery revascularization; renal artery stenosis (refers to diameter stenosis ≥50%).
The incidence rate of adverse events and serious adverse events | 1 month, 2 months, 3 months, 6 months after the operation
  The number of adverse events and serious adverse events
The incidence rate of device defects. | during the operation
  The number of occurrences of device defects

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Sun Yat-sen University （Sun Yat-sen Memorial Hospital）, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No